CLINICAL TRIAL: NCT06377436
Title: Prevenzione Della disabilità Nella Persona Anziana Fragile Attraverso un Innovativo Programma di Allenamento Personalizzato e Multidimensionale
Brief Title: Prevention of Disability in the Frail Elderly Person Through an Innovative Customised and Multidimensional Training Programme
Acronym: PRAISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof.ssa Gabriella Cerri, Full professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRAISE
Record Dates: First submitted 2024-03-21; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Frailty
Keywords: Frailty; cognitive function; elderly
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIVIDAT SENSO GROUP (Experimental): 40 frail subjects who will undergo the experimental training - "DIVIDAT SENSO training" on the Locomotor, Sensory and Cognitive domains. Traning wilk be performed at IRCCS Galeazzi-Sant'Ambrogio Hospital (5 non-consecutive sessions every 15 days, for 1 year)
  Interventions: Behavioral: Experimental training
- STANDARD OF CARE GROUP (No Intervention): 40 frail subjects will be subjected to good practice rules for all 5 domains of the intrinsic capacity. Subject will be followed for 1 year. No specific supervised training will be administered to this group.

INTERVENTIONS:
Behavioral: Experimental training — Through The Dividat Senso intelligent platform, subjects will be subjected to locomotion, cognitive and sensory domain-specific exercise programs. The exercises will be of increasing difficulty. Cognitive exercises will in fact be carried out by interacting with the DIVIDAT device consisting of a monitor and a pressure-sensitive platform through weight shifts, multidirectional steps and jumps.
  Arms: DIVIDAT SENSO GROUP

SUMMARY:
The goal of this clinical trial is to implement a personalized training program to prevent functional decline in frail subjects but not yet disable. The purpose of the project is to test the training in a subject at particularly high risk of entering the disabled condition. A total of 80 frail subjects, divide the participants into two groups "Divida Senso Group" (experimental group) and "Standard of care Group" (Control group) will be recruited.

The expected outcome is to slow down a functional decline not only in isolation in the domains trained by the program.

DETAILED DESCRIPTION:
INTRINSIC CAPACITY The "active and healthy" aging of each individual depends on the individual's "Intrinsic Capacity" (IC) and his or her interaction with the environment. Intrinsic Capacity is a composite index derived from the subject's assessment of 5 key domains on which the individual's perfect functionality is based. These domains are: Motricity (particularly locomotion), Sensory Competence (particularly referring to vision and hearing), Vitality (lifestyle), Cognitive Abilities, and Mood Status. The reduction in IC is physiological, but the rate at which the elderly person's functional reserve decreases can be variable, slower in some cases and faster in others, depending on various endogenous and environmental factors. Therefore, the elderly person is not inexorably destined for rapid decline as there is also a functional reserve in the aging organism.

CONSEQUENCES OF ISOLATION DUE TO THE COVID PANDEMIC The Covid pandemic produced very significant consequences especially for the elderly population. The isolation measures that were put in place during the pandemic highlighted, how much the drastic reduction in the ability to go out for common daily activities disrupted the lifestyle, reduced both motility and sociality of the elderly, possibly affecting the decline of intrinsic capacity. In addition, it was pointed out how lacking is the surveillance of the elderly in the area in terms of monitoring prevention and intervention.

THE FRAILTY CONDITION AND INDIVIDUAL AND SOCIAL CONSEQUENCES The rapid rate of decline in IC is very important as it can lead to frailty, a common geriatric condition characterized by extreme vulnerability of the body to stressors (endogenous and exogenous) with significantly increased risk of adverse health-related outcomes such as disability, institutionalization, hospitalization, and death. The consequences of frailty impair the individual's activity status and place a significant burden on the health care system. The annual health care cost per person in Europe can present a 3-fold increase depending on frailty status and care setting. However, frailty could potentially be reversible; its early detection should lead to the implementation of preventive strategies to correct abnormal deviations from the normal trajectory of aging by making the elderly population autonomous and active in society.

PURPOSE OF THE STUDY The project hypothesizes that frailty is caused by the subject's decline in IC, and thus can be considered a suitable model to test a training program targeting the domains of IC, with a focus on cognitive function, locomotion, and the sensory domain. The goal is to conduct a pilot study in frail elderly people in order to implement a personalized training program to prevent functional decline. The training will be conducted on a sensorized platform (DIVIDAT SENSO) capable of administering cognitive, motor, and dual task (integrated cognitive and motor) exercises. The purpose of the training is to improve the performance of the frail subject, and the evaluation of the training outcome will be done by comparing the results of the assessment battery at time T0, pre-training and T1 post-training. The DIVIDAT SENSO platform and all the instrumentation necessary for the assessment of the various performance domains of the subject are not the object of the study per se but a tool for its execution. An experimental population consisting of frail but not yet disabled individuals was chosen for the study. The choice of this condition for the study was based on the need to test the training in a subject at particularly high risk of entering the disabled condition (a so-called borderline subject, i.e., at the functional boundary between ability and disability) and losing independent living. The expected result is functional recovery not only in isolation in the domains trained by the program but, with a knock-on effect, on the others as well by going on to implement the entire IC. Significantly relevant results in this population would provide a solid scientific basis for the effectiveness of the program as it would affect a population already in very advanced stages of decline.

RELEVANCE AND PROSPECTS Having demonstrated the efficacy of training with the present project, it would be hoped to proceed with an extensive study on a larger population, over an extended study period, involving frail and non-frail subjects in order to verify the impact of training on the slope of physiological decline. Contextually, a network would be established to monitor the performance of the enrolled subjects, which transmitted to the primary care physician would allow active surveillance and the possibility of targeted intervention in case of pathological or borderline performance.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years,
* Fraiity index borderline based on the Searle scale (Searle et al.2008);
* Acceptance Agreement to take part in the study and signing of informed consent

Exclusion Criteria:

* Severe cognitive or motor deficits that make the patient unable to understand/fill out an informed consent or ambulate independently;
* Neurodegenerative disease affecting locomotor or sensorial system;
* Dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the Functional decline | through training completion, ( 1 year after training)
  Functional decline defined and measured by a reduction in ability to perform self-care activities of daily living (ADL) because of a decrement in physical or cognitive functioning or in 1 of 5 domains of intrinsic capacity (IC). Functional decline will be measured using Frailty Checklist (score range 0-18; 0=not frail- 18 Severe frailty) and Short Physical Performances Battery (SPPB; scores range from 0 = worst performance to 12 =best performance).
Intrinsic Capacity (IC) | through training completion, ( 1 year after training)
  Quantitative assessment of the five domains of the IC. Each domain will be measured using specific test.
  1. Cognition : Mini Mental State Examination (score range 0-30) , Fluency test, 15 Rey's words, H cancellation test (for the last three test the equivalent score is used - range 0=patological-4-better normal performance)
  2. Locomotion: Six minutes walking test, Timed Up and Go test (TUG) and cognitive TUG;
  3. Sensory: vision test and Whisper test for the hearing;
  4. Vitality: handgrip-strength and Mini Nutritional assessment.
  5. Psychological domain: Hospital Anxiety and Depression Scale (A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.)
  The interaction effect, among the 5 domains of the IC, will be measured using Spearman's rank correlation coefficient. This identifications it allows whether the intervention on specific domains of the IC will spread the favourable effect on others as well.
Intreaction between IC and cardiac autonomic control (CAC) | through training completion, ( 1 year after training)
  The association between IC and CAC (10 minutes ECG in rest and stand) . Application. Effect on CAC. This is indeed enhanced by interventions that can influence performance and individual functioning such as physical/mental training.

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriella CERRI, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakker J, Donath L, Rein R. Balance training monitoring and individual response during unstable vs. stable balance Exergaming in elderly adults: Findings from a randomized controlled trial. Exp Gerontol. 2020 Oct 1;139:111037. doi: 10.1016/j.exger.2020.111037. Epub 2020 Jul 28. PMID 32730797
- [Background] Carlesimo GA, Caltagirone C, Gainotti G. The Mental Deterioration Battery: normative data, diagnostic reliability and qualitative analyses of cognitive impairment. The Group for the Standardization of the Mental Deterioration Battery. Eur Neurol. 1996;36(6):378-84. doi: 10.1159/000117297. PMID 8954307
- [Background] Guyatt GH, Sullivan MJ, Thompson PJ, Fallen EL, Pugsley SO, Taylor DW, Berman LB. The 6-minute walk: a new measure of exercise capacity in patients with chronic heart failure. Can Med Assoc J. 1985 Apr 15;132(8):919-23. PMID 3978515
- [Background] Guigoz Y, Vellas B, Garry PJ. Assessing the nutritional status of the elderly: The Mini Nutritional Assessment as part of the geriatric evaluation. Nutr Rev. 1996 Jan;54(1 Pt 2):S59-65. doi: 10.1111/j.1753-4887.1996.tb03793.x. No abstract available. PMID 8919685
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Maguire, N., Prosser, S., Boland, R., & McDonnell, A. (1998). Screening for hearing loss in general practice using a questionnaire and the whisper test. The European Journal of General Practice, 4(1), 18-21.
- [Background] Gordon, W.A., Ruckdeschel-Hibbard, M., Egelko, S., Diller, L., Simmens, S., Langer, K. (1984). Single Letter Cancellation Test in Evaluation of the Deficits Associated with Right Brain Damage: Normative Data on the Institute of Rehabilitation Medicine Test Battery. New York: New York University Medical Center
- [Background] Novelli, P., Capitani, L., Vallar, C., & Cappa, S. (1986). Test di fluenza verbale. Archivio di Psicologia, Neurologia e Psichiatria, 47(4), 477-506.
- [Background] Pavey TG, Gomersall SR, Clark BK, Brown WJ. The validity of the GENEActiv wrist-worn accelerometer for measuring adult sedentary time in free living. J Sci Med Sport. 2016 May;19(5):395-9. doi: 10.1016/j.jsams.2015.04.007. Epub 2015 Apr 17. PMID 25956687
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Searle SD, Mitnitski A, Gahbauer EA, Gill TM, Rockwood K. A standard procedure for creating a frailty index. BMC Geriatr. 2008 Sep 30;8:24. doi: 10.1186/1471-2318-8-24. PMID 18826625
- [Background] Tombaugh TN, McIntyre NJ. The mini-mental state examination: a comprehensive review. J Am Geriatr Soc. 1992 Sep;40(9):922-35. doi: 10.1111/j.1532-5415.1992.tb01992.x. PMID 1512391
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Bailey IL, Lovie JE. New design principles for visual acuity letter charts. Am J Optom Physiol Opt. 1976 Nov;53(11):740-5. doi: 10.1097/00006324-197611000-00006. PMID 998716